CLINICAL TRIAL: NCT05625971
Title: Non-Invasive Minimal Residual Disease (MRD) Assessment in Multiple Myeloma Via Functional Imaging and Liquid Biopsy
Brief Title: Non-invasive MRD Assessment in Multiple Myeloma
Acronym: NIRVANA
Status: Completed | Type: Observational
Sponsor: Rajshekhar Chakraborty, MD (Other)
Collaborators: Hope Foundation (Other)
Responsible Party: Sponsor-Investigator, Rajshekhar Chakraborty, MD, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Other Study IDs: AAAU0686
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Myeloma
Keywords: Liquid biopsy; Minimal Residual Disease (MRD); Functional imaging
MeSH Terms: conditions — Neoplasms, Plasma Cell; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone marrow aspirate and biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Myeloma Group: Patients with newly diagnosed and previously treated multiple myeloma will receive bone marrow sampling and functional imaging.
  Interventions: Other: MRD Assessment

INTERVENTIONS:
Other: MRD Assessment — MRD assessment includes liquid biopsy and functional imaging. Liquid biopsy will be performed by the Adaptive ClonoSEQ® assay in peripheral blood. Functional imaging will be performed by whole body diffusion-weighted magnetic resonance imaging (WB-DWI).

SUMMARY:
The purpose of this study is to investigate the sensitivity and accuracy of non-invasive MRD assessment using liquid biopsy (blood draw) and functional imaging (whole body MRI) in participants with new diagnosed and previously treated multiple myeloma. The long-term goal of this study is to investigate whether non-invasive methods for MRD assessment can replace bone marrow aspiration and biopsy in a substantial percentage of participants with multiple myeloma.

DETAILED DESCRIPTION:
There is an unmet clinical need for an easier, non-invasive, and reliable method to perform MRD assessments that can be used in clinical trials and routine practice. The two non-invasive modalities that are most promising for MRD assessment are liquid biopsy to detect circulating tumor cells (CTCs) and functional imaging to detect focal myeloma lesions. However, there are no prospective data on the sensitivity and specificity of non-invasive MRD assessment with respect to the gold standard of bone marrow sampling.

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥18 years
* Patients with newly diagnosed multiple myeloma
* Patients with previously treated multiple myeloma with a maximum of two prior lines of therapy
* Expected life expectancy of greater than one year and intention to start a new line of treatment

Exclusion Criteria:

* Patients without cognitive capacity to give informed consent for participation
* Patients with contraindications to MRI, which include the following:
* Claustrophobia, which, at investigator's discretion, would prohibit patient from undergoing whole body diffusion-weighted magnetic resonance imaging (WB-DWI)
* Pacemaker
* Metallic implants, which would prohibit patient from undergoing MRI All subjects will be screened for any contraindication to MRI as per their guidelines at the time of patient enrollment.
* Patients must not receive granulocyte colony stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) injection within 1 week prior to WB-DWI.
* Patients must not have been initiated on treatment prior to baseline disease assessment by bone marrow aspiration/biopsy and/or WB-DWI Up to 160 mg of dexamethasone (or equivalent) and/or 1 dose of bortezomib (+/- Cyclophosphamide-Dexamethasone) is allowed prior to disease assessment by bone marrow aspiration and WB-DWI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed or previously treated myeloma who are initiating a new line of therapy will be recruited.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity of non-invasive MRD assessment | 6 months
  MRD assessment includes liquid biopsy and functional imaging.
Specificity of non-invasive MRD assessment | 6 months
  MRD assessment includes liquid biopsy and functional imaging.

SECONDARY OUTCOMES:
Sensitivity of two MRD-testing algorithms | 6 months
  Combining liquid biopsy, functional imaging, and bone marrow sampling against the reference of bone marrow sampling in patients
Specificity of two MRD-testing algorithms | 6 months
  Combining liquid biopsy, functional imaging, and bone marrow sampling against the reference of bone marrow sampling in patients
Progression Free Survival | 2 years
  The progression-free survival (PFS) will be calculated of patients who are MRD-positive and MRD-negative on each modality (liquid biopsy, functional imaging, and bone marrow sampling)
Overall Survival | 2 years
  The overall survival (OS) will be calculated of patients who are MRD-positive and MRD-negative on each modality (liquid biopsy, functional imaging, and bone marrow sampling)

CONTACTS AND LOCATIONS:
Overall Officials: Chakraborty Chakraborty, MD, Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian Hospital/Columbia University Irving Medical Center, New York, New York, United States